CLINICAL TRIAL: NCT01977066
Title: SUPPORT - Study Supervised Progressive Resistance Training for Pancreatic Cancer Patients: a Randomized Controlled Intervention Trial
Brief Title: Exercise Intervention Study for Pancreatic Cancer Patients
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University of Heidelberg Medical Center (Other); Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SUPPORT
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; exercise training; quality of life; physical functioning
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Six months supervised exercise training (Experimental)
  Interventions: Behavioral: Six months supervised resistance training
- Six months home-based exercise training (Experimental)
  Interventions: Behavioral: Six months home-based exercise training
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Six months supervised resistance training — progressive resistance training (2x/week), starting at the earliest 8 weeks after surgery until maximum 12 months after the surgery with only low-to-moderate-intensity training during the first 4 weeks.
  Arms: Six months supervised exercise training
Behavioral: Six months home-based exercise training — Home-based exercise training (2x/week) with initial counseling and weekly telephone contact starting at the earliest 8 weeks after surgery until maximum 12 months after the surgery.
  Arms: Six months home-based exercise training

SUMMARY:
The purpose of this study is to compare the effects of two specific exercise interventions and one standard care control arm on physical functioning.The investigators expect that supervised training is most beneficial to the patients. However, they also expect some benefit for patients in the home-based training.

DETAILED DESCRIPTION:
The randomized-controlled balanced-parallel-group trial included 65 adult pancreatic cancer patients (stage I-IV) from the University Surgery Clinic in Heidelberg. The study compared two specific exercise interventions and one standard care control arm. The intervention programs were (1) a 6-month supervised moderate-to-high-intensity, progressive resistance training, and (2) a 6-month home-based exercise training. Thus, the two interventions differed primarily by the intensity and mode-of-administration of the intervention. Both interventions started at the earliest 8 weeks after surgery to allow for wound healing until Maximum 12 months after the surgery. The supervised progressive training started with only moderate-intensity training during the first 4 weeks. Only patients without comorbidities that preclude participation in the intervention arms (e.g. severe pain, heart insufficiency, reduced standing or walking ability) were eligible.

The primary objective is to compare the effects of the different interventions on physical functioning, measured as change from baseline to 6 months. Additional endpoints are overall quality of life, fatigue, endurance, and strength performance, adherence to the interventions, discontinuation of adjuvant therapy, body weight and composition, disease progression, overall and progression-free survival. All outcomes has been assessed every 3 months for a minimum follow-up period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer patients (stage I-IV)
* Patients ≥ 18 years of age
* Resection performed at the University Clinic of Heidelberg
* Sufficient German language skills
* Signed informed consent

Exclusion Criteria:

• Presence of comorbidities that preclude participation in the intervention arms (e.g. severe pain, heart insufficiency, reduced standing or walking ability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Physical functioning score, as assessed by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) EORTC QLQ-C30 | Change from baseline to end of intervention (after 6 months)

SECONDARY OUTCOMES:
Overall quality of life from EORTC QLQ-C30 and the specific module for pancreatic cancer(QLQ-PAN26) | change from Baseline to end of intervention (6 months)

OTHER OUTCOMES:
Fatigue (Multidimensional Fatigue Inventory (MFI)) | change from baseline to end of intervention (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Karen G Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center (DKFZ)/ German National Center for Tumor Diseases (NCT)
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939
- [Derived] Wochner R, Clauss D, Nattenmuller J, Tjaden C, Bruckner T, Kauczor HU, Hackert T, Wiskemann J, Steindorf K. Impact of progressive resistance training on CT quantified muscle and adipose tissue compartments in pancreatic cancer patients. PLoS One. 2020 Nov 30;15(11):e0242785. doi: 10.1371/journal.pone.0242785. eCollection 2020. PMID 33253318
- [Derived] Wiskemann J, Clauss D, Tjaden C, Hackert T, Schneider L, Ulrich CM, Steindorf K. Progressive Resistance Training to Impact Physical Fitness and Body Weight in Pancreatic Cancer Patients: A Randomized Controlled Trial. Pancreas. 2019 Feb;48(2):257-266. doi: 10.1097/MPA.0000000000001221. PMID 30589829